- **Protocol number:** MTI-107
- **Document title:** An open-label long-term safety study of serlopitant for the treatment of pruritus.
- Version numbers: SAP Version 4.0
  Date of the documents: 12 May 2020
- **NCT number:** NCT03540160

# STATISTICAL ANALYSIS PLAN

Cto. do. Title.

Study Title: AN OPEN-LABEL LONG-TERM SAFETY

MTI-107

STUDY OF SERLOPITANT FOR THE

TREATMENT OF PRURITUS

Development Phase of Study: Phase 3

Sponsor: Menlo Therapeutics Inc.

200 Cardinal Way, 2<sup>nd</sup> Floor Redwood City, CA 94063

**USA** 

Sponsor Contact:

Statistical Analysis Plan based on

Protocol Version:

Protocol Number:

Version 3.0, 21 March 2019

Statistical Analysis Plan Date: 12 May 2020 Statistical Analysis Plan Version: Version 4

Confidentiality Statement:

This document is a confidential communication of Menlo Therapeutics Inc. As such, the recipients agree not to disclose or reproduce, without prior written approval, this document and any attachments, except to appropriate Institutional Review Boards, Ethics Committees, representatives of the US Food and Drug Administration, other regulatory agencies or as otherwise required by applicable laws or regulations.

Statistical Analysis Plan for Menlo Therapeutics Inc. Protocol Number: MTI-107

| Authored by: | |
|--------------|-----|
| | PPD |

# TABLE OF CONTENTS

| 1. | LIS | T OF A | ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | INT | RODU | UCTION | 6 |
| 3. | STU | J <b>DY O</b> | BJECTIVES | 6 |
| 4. | STUDY DESIGN | | | 7 |
| | 4.1 | Overa | ll Study Design | 7 |
| | | 4.1.1 | Schedule of Visits and Assessments | 7 |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | 7 |
| | | 4.1.3 | Blinding | 7 |
| 5. | EFI | FICAC | Y AND SAFETY ENDPOINTS | 7 |
| | 5.1 | Effica | cy Endpoints | 7 |
| | 5.2 | Safety | Endpoints | 8 |
| 6. | STA | ATISTI | ICAL AND ANALYTICAL PLANS | 8 |
| | 6.1 | Gener | al Methodology | 8 |
| | | 6.1.1 | Statistical Analysis | 8 |
| | | 6.1.2 | Baseline Definition | 8 |
| | | 6.1.3 | Visit Windowing | 9 |
| | | 6.1.4 | Adjustments for Covariates | 9 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | |
| | | 6.1.6 | Multicenter Studies | 9 |
| | | 6.1.7 | Multiple Comparisons/Multiplicity | 9 |
| | | 6.1.8 | Examination of Subgroups | 9 |
| | 6.2 | Dispo | sition of Subjects | 9 |
| 6.3 Protocol Deviations | | col Deviations | 9 | |
| | 6.4 | Data S | Sets Analyzed | 10 |
| | | 6.4.1 | Safety Population | 10 |
| 6.5 Demographic and Other Baseline Characteristics | | 10 | | |
| | 6.6 Prior and Concomitant Medications | | 10 | |
| 6.7 Analysis of Efficacy | | rsis of Efficacy | 10 | |
| | 6.8 | Safety | Evaluation | 10 |
| | | 6.8.1 | Extent of Exposure | 10 |
| | | 6.8.2 | Adverse Events | 10 |
| | | 6.8.3 | Clinical Laboratory Evaluation | 11 |
| | | 6.8.4 | Other Observations Related to Safety | 11 |
| | | | 6.8.4.1 Electrocardiogram Measurements | 11 |

| | 6.8.4.2 | Vital Signs | 11 |
|---|---|---|---|
| | 6.8.4.3 | Physical Exams | 11 |
| | 6.8.4.4 | Menstrual Diaries | 11 |
| | 6.8.4.5 | Hospital Anxiety and Depression Scale (HADS) | 11 |
| | 6.8.4.6 | Epworth Sleepiness Scale (ESS) | 11 |
| 7. | <b>DETERMINATION</b> | OF SAMPLE SIZE | 12 |
| 8. | CHANGES IN THE I | PLANNED ANALYSES | 12 |
| 9. | INDEX OF PLANNE | D END-OF-TEXT TABLES AND FIGURES | 13 |
| 10. | INDEX OF PLANNE | D LISTINGS | 27 |

# **Revision History:**

| Version | Date | Summary of Changes | Author |
|---|---|---|---|
| Version 1 | 13 November 2018 | Original document | PPD |
| Version 2 | 03 April 2019 | Updated title page to reflect current version of protocol. Updated SAP version and date. | PPD |
| | | Updated Section 7 to include expected number of subjects to be enrolled. | |
| Version 3 | 11 February 2020 | Updated SAP version and date. | PPD |
| | | Editorial and grammatical updates including abbreviations and references. | |
| | | Added table, figure and listing shells. | |
| Version 4 | 12 May 2020 | Updated SAP version and date. | PPD |
| | | Updated SAP throughout, including text, table shells and listing shells to facilitate abbreviated study report. | |

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AD Atopic Dermatitis
AE(s) Adverse event(s)

DLQI Dermatology Life Quality Index

ECG Electrocardiogram
EOS End of Study
EOT End of Treatment

ESS Epworth Sleepiness Scale

HADS Hospital Anxiety and Depression Scale

IGA PN-S Investigator's Global Assessment of Prurigo Nodularis Stage

MedDRA Medical Dictionary for Regulatory Activities

PN Prurigo Nodularis

SAE(s) Serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

TEAE(s) Treatment-emergent adverse event(s)

WHO-DD World Health Organization Drug Dictionary

WI-NRS Worst-Itch Numeric Rating Scale

#### 2. INTRODUCTION

The MTI-107 study described herein is an open-label study to assess the long-term safety of serlopitant in adults with pruritus associated with prurigo nodularis (PN), atopic dermatitis (AD), or psoriasis.

Subjects enrolled in MTI-107 may have or may not have participated in previous Menlo Therapeutics Inc. studies. Previous study participation includes studies in PN (MTI-105, MTI-106, TCP-102), in AD (MTI-103) and in psoriasis (MTI-109).

The MTI-107 study has been terminated early by Sponsor. The Statistical Analysis Plan has been updated to facilitate an abbreviated clinical study report.

#### 3. STUDY OBJECTIVES

The primary objective of this study is to assess the long-term safety of serlopitant in adults with pruritus associated with PN, AD, or psoriasis.

The secondary objectives of this study are to assess the change in severity of pruritus in subjects with PN, AD, or psoriasis using the worst-itch numeric rating scale (WI-NRS); to assess the change in severity and extent of PN using the Investigator's Global Assessment of PN Stage

Statistical Analysis Plan for Menlo Therapeutics Inc. Protocol Number: MTI-107

(IGA PN-S), for those subjects with PN; and to assess whether serlopitant produces physical dependence.

#### 4. STUDY DESIGN

# 4.1 Overall Study Design

This is a multicenter, open-label study to assess the long-term safety of serlopitant in adults with pruritus associated with PN, AD, or psoriasis. Eligible subjects who have completed selected studies of serlopitant may be given the opportunity, at the Investigator's discretion, to consent to and participate in this open-label study, regardless of their treatment allocation in prior studies. If deemed necessary by Menlo Therapeutics to meet enrollment objectives, eligible subjects who have not participated in a prior serlopitant study may also be enrolled in study MTI-107. Approximately 120 study sites may enroll subjects in this long-term safety study.

This study will consist of two periods, for a total study period of 57 weeks:

• Treatment period: 52 weeks

• Post-drug observation period: 5 weeks

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 6.4 and Appendix A of the Protocol.

# 4.1.2 Method of Assigning Subjects to Treatment Groups

This is an open-label single-arm study. Eligible subjects will receive serlopitant 5 mg tablets.

# 4.1.3 Blinding

This is an open-label study.

#### 5. EFFICACY AND SAFETY ENDPOINTS

# 5.1 Efficacy Endpoints

Efficacy endpoints are as follows:

- Change from baseline in WI-NRS to Weeks 4, 8, 20, 28, 36, 44, and 52
- Change from baseline in Dermatology Life Quality Index (DLQI) to Weeks 20, 36, and
   52
- Change from baseline in Investigator's Global Assessment of PN Stage (IGA PN-S) to Weeks 4, 8, 20, 28, 36, 44, and 52

# 5.2 Safety Endpoints

Safety endpoints include the following:

- Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
- Changes from baseline in clinical laboratory parameters
- Changes from baseline in vital sign and electrocardiogram (ECG) parameters
- Change from baseline in the Hospital Anxiety and Depression Scale (HADS)
- Change from baseline in the Epworth Sleepiness Scale (ESS)
- Assessment of physical dependence following chronic study drug exposure, in the monitored 5-week post-drug discontinuation period

#### 6. STATISTICAL AND ANALYTICAL PLANS

# 6.1 General Methodology

All statistical processing will be performed using SAS® Version 9.3 or later, unless otherwise stated. No interim analyses are planned. Endpoints will be summarized with descriptive statistics by visit. For continuous variables, the following information will be presented: n (number of subjects), mean, standard deviation (SD), median, minimum and maximum. For categorical variables, counts and percentages will be presented.

Reported adverse events (AEs), medical history, and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology. Concomitant medications will be classified on the basis of World Health Organization Drug Dictionary (WHO-DD) terminology.

# 6.1.1 Statistical Analysis

All summary tables and data listings will be prepared by QST Consultations, Ltd., utilizing SAS® Version 9.3 or later software.

The standard operating procedures of QST Consultations, Ltd. will be followed in the creation and quality control of all data displays.

#### **6.1.2** Baseline Definition

No change from baseline summaries will be created.

# 6.1.3 Visit Windowing

Data will be provided in by-subject listings based on nominal visit indications.

# 6.1.4 Adjustments for Covariates

No inferential statistical analyses are planned.

### 6.1.5 Handling of Dropouts or Missing Data

Summary statistics will generally be reported based upon observed data. Should a determination of treatment period (on treatment, pre-treatment, post-treatment) be required for AEs or concomitant medication but the corresponding date is missing, or is a partial date, the event/medication will be considered on treatment unless the portions of the date that are available indicate this is not possible.

#### **6.1.6** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling all the data for summaries. Every effort will be made to promote consistency in study execution at each study site.

# 6.1.7 Multiple Comparisons/Multiplicity

No inferential statistical analyses are planned.

# **6.1.8** Examination of Subgroups

No subgroup summaries will be created.

# 6.2 Disposition of Subjects

An accounting of all enrolled subjects by disposition will be presented. Subjects who discontinue study drug prematurely or withdraw from the study will be summarized and listed, with a description of the reason for early termination/withdrawal.

The number of subjects included in the safety population will be summarized. Subjects who are excluded from the safety population will be summarized by the reasons for exclusion.

#### **6.3** Protocol Deviations

Protocol deviations will be presented in a data listing.

# 6.4 Data Sets Analyzed

# 6.4.1 Safety Population

All subjects who receive at least 1 confirmed dose of study drug and have at least 1 post-baseline safety assessment or a reported TEAE will be included in the safety population. All analyses will be performed using the safety population.

# 6.5 Demographic and Other Baseline Characteristics

Sex, race, and ethnicity will be summarized by counts and percentages. Age, height (cm), and weight (kg) will be summarized with descriptive statistics.

Medical histories will be coded using MedDRA and presented in a by-subject listing.

Disease history (PN, AD, psoriasis) will be presented in a by-subject listing.

#### 6.6 Prior and Concomitant Medications

Prior and concomitant medications will be coded by the WHO-DD to Anatomical Therapeutic Classification (ATC) and preferred drug name.

A by-subject listing of all prior and concomitant medications will be presented. The associated by-subject listing will have a prior/concomitant determination that is based on the date of first dose.

# 6.7 Analysis of Efficacy

Efficacy data will be provided in by-subject listings.

# **6.8** Safety Evaluation

# **6.8.1** Extent of Exposure

The extent of exposure to study drug will be summarized by days with exposure and total number of tablets used. Subjects will be considered having 6-Month exposure if the date of first dose – date of last dose + 1 is greater than or equal to 182 days. Subjects will be considered having 1-Year exposure if date of first dose – date of last dose + 1 is greater than or equal to 358 days, considering the allowable -7 day window for the Week 52 visit.

#### 6.8.2 Adverse Events

All AEs will be classified by system organ class and preferred term using the MedDRA. TEAEs will be tabulated in a manner which provides information about the incidence of TEAEs for the entire study. For incidence reporting, if a subject reported more than one TEAE that was coded to the same system organ class or preferred term, the subject will be counted only once for that

specific system organ class or preferred term. An overview of AEs, which includes subject incidence of AEs, TEAEs, treatment-related TEAEs, TEAEs by severity, SAEs, deaths, and AEs leading to discontinuation of study drug, will be presented.

All information pertaining to AEs noted during the study will be listed by subject and will include a verbatim description of the event as reported by the investigator, as well as the preferred term, system organ class, start date, end date (if ended), seriousness, severity, action taken regarding the study drug, outcome, and relationship to the study drug. In addition, a listing of subjects who prematurely discontinued study drug due to AEs will be provided.

SAEs will be listed and summarized in a similar manner to AEs.

# 6.8.3 Clinical Laboratory Evaluation

By-subject listings of all laboratory data, as well as abnormal laboratory results, will be presented. Clinically significant laboratory results will be recorded as an AE.

# **6.8.4** Other Observations Related to Safety

# **6.8.4.1 Electrocardiogram Measurements**

Data will be provided in a by-subject listing.

# 6.8.4.2 Vital Signs

Data will be provided in a by-subject listing.

# 6.8.4.3 Physical Exams

Clinically significant physical exam findings will be recorded by the sites within medical history or adverse events and otherwise not summarized. Data will be provided in a by-subject listing.

#### **6.8.4.4 Menstrual Diaries**

Data will be provided in a by-subject listing.

# 6.8.4.5 Hospital Anxiety and Depression Scale (HADS)

Data will be provided in a by-subject listing.

# 6.8.4.6 Epworth Sleepiness Scale (ESS)

Data will be provided in a by-subject listing.

# 7. DETERMINATION OF SAMPLE SIZE

No formal sample size calculations were performed. Up to 700 adult subjects with pruritus associated with PN, AD, or psoriasis will be enrolled in this study.

# 8. CHANGES IN THE PLANNED ANALYSES

No graphs of laboratory values over time will be created.

Planned analyses have been updated to facilitate an abbreviated clinical study report.

# 9. INDEX OF PLANNED END-OF-TEXT TABLES AND FIGURES

| Table 14.0.1.1: Summar | ry of Subject Completion/Discontinuation (Enrolled Subjects) | 14 |
|---|---|---|
| Table 14.0.2.1: Summar | ry of Subjects Excluded from Analyses (Enrolled Subjects) | 15 |
| Table 14.1.1.1: Summar | ry of Subject Demographics (Safety Population) | 16 |
| Table 14.3.0.1: Summar | ry of Extent of Exposure (Safety Population) | 18 |
| Table 14.3.1.1.1: Ove | rall Summary of Treatment-Emergent Adverse Events (TEAEs) (Sa Population) | _ |
| Table 14.3.1.1.2.1: Sum | nmary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Sepulation) | Safety<br>20 |
| Table 14.3.1.1.3.1: Sum | nmary of Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug (Safety Population) | 21 |
| Table 14.3.1.1.4.1: Sum | nmary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population) | 22 |
| Table 14.3.1.1.5.1: Sum | nmary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population) | 23 |
| Table 14.3.1.3.1.1: Sum | Events (TEAEs) by MedDRA System Organ Class and Preferred (Safety Population) | Term<br>24 |
| Table 14.3.1.3.2.1: Sum | nmary of Subjects Reporting Serious Treatment-Emergent Adverse<br>Events (TEAEs) by Severity (Safety Population) | 25 |
| Table 14.3.1.3.3.1: Sum | nmary of Subjects Reporting Serious Treatment-Emergent Adverse<br>Events (TEAEs) by Relationship to Study Drug (Safety Population | n)26 |

Statistical Analysis Plan for Menlo Therapeutics Inc. Protocol Number: MTI-107

Table 14.0.1.1: Summary of Subject Completion/Discontinuation (Enrolled Subjects)

| | Serlopitant 5 mg |
|-------------------------------------------|------------------|
| | (N=xxx) |
| Completed Treatment | |
| Yes | xx ( xx.x%) |
| No | xx ( xx.x%) |
| Reason for Discontinuation from Treatment | |
| Adverse Event | xx (xx.x%) |
| Lack of Efficacy | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) |
| Investigator Decision | xx ( xx.x%) |
| Withdrawal by Subject from Treatment | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) |
| Sponsor Decision | xx ( xx.x%) |
| Other | xx ( xx.x%) |
| Completed Follow-up | |
| Yes | xx ( xx.x%) |
| No | xx ( xx.x%) |
| Reason for Discontinuation from Follow-up | |
| Withdrawal by Subject from Study | xx ( xx.x%) |
| Lost to Follow-up | $xx(x^0/x)$ |
| Other | XX (XX.X%) |

Table 14.0.2.1: Summary of Subjects Excluded from Analyses (Enrolled Subjects)

| | Serlopitant 5 mg (N=xxx) |
|----------------------------------|--------------------------|
| Safety Population | (14-AAA) |
| Number of Subjects Included | xx ( xx.x%) |
| Number of Subjects Excluded | XX (XX,X%) |
| Reason for Exclusion | |
| No Evidence of Subject Dosing | XX (XX,X%) |
| No Post-Baseline Assessment/TEAE | XX (XX,X%) |

Table 14.1.1.1: Summary of Subject Demographics (Safety Population)
(Page 1 of 2)

| | Serlopitant 5 mg |
|---|---|
| | (N=xxx) |
| Age (years) | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Sex | |
| n | XXX |
| Male | xx ( xx.x%) |
| Female | xx ( xx.x%) |
| Ethnicity | |
| n | XXX |
| Hispanic or Latino | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) |
| Race | |
| n | XXX |
| American Indian or Alaska Native | xx ( xx.x%) |
| Asian | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ |
| Black or African American | XX (XX.X%) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X%) |
| White | XX (XX,X'') |
| Multiple/Other | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ |
| manple, outer | AA ( AA.A./0) |

Table 14.1.1.1: Summary of Subject Demographics (Safety Population)
(Page 2 of 2)

| | Serlopitant 5 mg (N=xxx) |
|--------------|--------------------------|
| Height (cm) | (IV AAA) |
| N | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Weight (kg) | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

Table 14.3.0.1: Summary of Extent of Exposure (Safety Population)

| | Serlopitant 5 mg (N=xxx) |
|---------------------------------------------|--------------------------|
| otal Number of Tablets Used | XXX |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| otal Number of Days of Exposure | XXX |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Subjects with 6-Month Exposure <sup>a</sup> | xx ( xx.x%) |
| Subjects with 1-Year Exposure <sup>a</sup> | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Subjects considered having 6-Month exposure if date of first dose – date of last dose + 1 is greater than or equal to 182 days.

Subjects considered having 1-Year exposure if date of first dose – date of last dose + 1 is greater than or equal to 358 days, considering the allowable -7 day window for the Week 52 visit.

Table 14.3.1.1.1: Overall Summary of Treatment-Emergent Adverse Events (TEAEs) (Safety Population)

| | Serlopitant 5 mg |
|---|---|
| | (N=xxx) |
| Subjects with any TEAE | XX ( XX.X%) |
| Number of TEAEs | XXX |
| Subjects with any Related TEAE | xx ( xx.x%) |
| Number of Related TEAEs | XXX |
| Subjects with any Serious TEAE | xx ( xx.x%) |
| Number of Serious TEAEs | XXX |
| Subjects with any Related Serious TEAE | xx ( xx.x%) |
| Number of Related Serious TEAEs | XXX |
| Subjects who Died | xx ( xx.x%) |
| Subjects who Discontinued Study Drug Due to TEAE | xx ( xx.x%) |
| Maximum Severity by Subject | |
| Grade 5 | $XX \left( XX.X^{0}/_{0} \right)$ |
| Grade 4 | xx (xx.x%) |
| Grade 3 | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) |
| Maximum Relationship by Subject | |
| Likely Related | xx ( xx.x%) |
| Likely Unrelated | xx ( xx.x%) |

Table 14.3.1.1.2.1: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|---|---|
| Total | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

MedDRA Version 21.1.

Table 14.3.1.1.3.1: Summary of Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|---|---|
| Total | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

MedDRA Version 21.1.

Table 14.3.1.1.4.1: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|------------------------------------------------|--------------------------|
| Total | |
| Grade 5 | xx (xx.x%) |
| Grade 4 | xx (xx.x%) |
| Grade 3 | xx (xx.x%) |
| Grade 2 | xx (xx.x%) |
| Grade 1 | xx ( xx.x%) |
| System Organ Class | |
| Grade 5 | xx (xx.x%) |
| Grade 4 | xx (xx.x%) |
| Grade 3 | xx (xx.x%) |
| Grade 2 | xx (xx.x%) |
| Grade 1 | xx ( xx.x%) |
| Preferred Term | |
| Grade 5 | xx ( xx.x%) |
| Grade 4 | xx (xx.x%) |
| Grade 3 | xx (xx.x%) |
| Grade 2 | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

MedDRA Version 21.1.

Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Life Threatening; Grade 5=Death.

Table 14.3.1.1.5.1: Summary of Subjects Reporting Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug
(Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|---|---|
| Total<br>Likely Related<br>Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |
| System Organ Class Likely Related Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term Likely Related Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

MedDRA Version 21.1.

# Table 14.3.1.3.1.1: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term (Safety Population) (Page 1 of xx)

| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|---|---|
| Total | xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: TEAEs are AEs with an onset date after first dose of study drug.

MedDRA Version 21.1.

Table 14.3.1.3.2.1: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Severity (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|------------------------------------------------|--------------------------|
| Total | |
| Grade 5 | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) |
| System Organ Class | |
| Grade 5 | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) |
| Preferred Term | |
| Grade 5 | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) |
| Grade 3 | xx ( xx,x%) |
| Grade 2 | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

MedDRA Version 21.1.

Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Life Threatening; Grade 5=Death.

Table 14.3.1.3.3.1: Summary of Subjects Reporting Serious Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Drug (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Serlopitant 5 mg (N=xxx) |
|---|---|
| Total Likely Related Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |
| System Organ Class<br>Likely Related<br>Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term Likely Related Likely Unrelated | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more TEAEs that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

MedDRA Version 21.1.

# 10. INDEX OF PLANNED LISTINGS

| Listing 16.2.1.1: Subject Disposition Information | 29 |
|---|---|
| Listing 16.2.1.2: Discontinued Subjects | 30 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Not Met | 31 |
| Listing 16.2.3: Analysis Populations | 32 |
| Listing 16.2.4.1: Subject Demographic Information | 33 |
| Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms | 34 |
| Listing 16.2.4.2.2: Medical History | 35 |
| Listing 16.2.4.3: Pruritic Disease History | 36 |
| Listing 16.2.4.4.1: Unique Medication Names Coded to WHO DDE ATC Level 2 Terms and Preferred Names | 37 |
| Listing 16.2.4.4.2: Concomitant Medications | 38 |
| Listing 16.2.4.5: Concomitant Procedures/Therapies | 39 |
| Listing 16.2.4.6: Physical Examination | 40 |
| Listing 16.2.5.1: Study Visit Compliance | 41 |
| Listing 16.2.5.2: Study Drug Dispensing and Return | 42 |
| Listing 16.2.6.1: Worst Itch Numeric Rating Scale (WI-NRS) | 43 |
| Listing 16.2.6.2: IGA PN-S Results. | 44 |
| Listing 16.2.6.3: Dermatology Life Quality Index (DLQI) | 45 |
| Listing 16.2.6.4: Photography | 46 |
| Listing 16.2.7.1.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | 47 |
| Listing 16.2.7.1.2: Treatment-Emergent Adverse Events | 48 |
| Listing 16.2.7.1.3: Serious Adverse Events | 49 |
| Listing 16.2.7.1.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events | 50 |
| Listing 16.2.7.2.1: Hospital Anxiety and Depression Scale | 51 |
| Listing 16.2.7.2.2: Epworth Sleepiness Scale | 52 |
| Listing 16.2.7.3: Menstrual Diary | 53 |
| Listing 16.2.8.1: Pregnancy Test Results | 54 |
| Listing 16.2.8.2.1: Laboratory Test Results. | 55 |
| Listing 16.2.8.2.2: Out of Range Laboratory Results | 56 |

| Listing 16.2.8.2.3: Laboratory Information Captured within Case Report Forms | 57 |
|---|---|
| Listing 16.2.8.2.4: Common Laboratory Comments Including Reference Ranges for Specific | <b>-</b> c |
| Laboratory Tests | 58 |
| Listing 16.2.8.3: Electrocardiogram Test Results | 59 |
| Listing 16.2.8.4: Vital Signs | 60 |

#### Listing 16.2.1.1: Subject Disposition Information (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date of Last Dose | R: Reason for Treatment Discontinuation P: Primary AE Number/Specify | E: Follow-up Discontinuation<br>Date (Day) <sup>1</sup><br>R: Reason for Follow-up<br>Discontinuation | D: Date of Last Contact P: Primary AE Number/Specify |
|---|---|---|---|---|
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxxxxxx xx xxxxxxxxx | D: xxxx-xx-xx<br>P: xxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx)<br>R: xxxxxxxxx xx xxxxxxxxx | D: xxxx-xx-xx<br>P: xxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx | R: xxxxxxxxx xxxx xxxxxxx xxxxx<br>P: xxxxxxxxxx | E: xxxx-xx-xx (xx)<br>R: xxxx xx xxxxxxxx | D:<br>P: xxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

#### Listing sorted by Subject.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose. Note: S = Safety Population.

# Listing 16.2.1.2: Discontinued Subjects (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date of Last Dose | R: Reason for Treatment Discontinuation P: Primary AE Number/Specify | E: Follow-up Discontinuation Date (Day)¹ R: Reason for Follow-up Discontinuation | D: Date of Last Contact<br>P: Primary AE Number/Specify |
|---|---|---|---|---|
| : xxxxxx | F: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxx | E: xxxx-xx-xx (xx) | D: xxxx-xx-xx |
| : XXXX | L: xxxx-xx-xx | P: xxxxxxxxx | R: XXXXXXXXXX XX XXXXXXXXX | P: xxxxxxxxxx |
| : xxxxxxxxx | _, | | | |
| : xxxxxx | F: xxxx-xx-xx | R: xxxxxxxxx xx xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | D: xxxx-xx-xx |
| : xxxx | L: xxxx-xx-xx | P: xxxxxxxxxx | R: xxxxxxxxx xx xxxxxxxxx | P: xxxxxxxxxx |
| : xxxxxxxxx | | | | |
| S: xxxxxx | F: xxxx-xx-xx | R: xxxxxxxx xxxx xxxxxxx xxxxx | E: xxxx-xx-xx (xx) | D: |
| A: xxxx | L: xxxx-xx-xx | P: xxxxxxxxx | R: xxxx xx xxxxxxxx | P: xxxxxxxxxx |
| : xxxxxxxxx | | | | |

Listing sorted by Subject.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.2.1: Inclusion/Exclusion Criteria Not Met (Page xx of yy)

| Subject | Age/Sex | Evaluable | Criterion Failed | Description |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx xxx xx xxxxxx xxxx xxxx xxxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** ************* |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxx | xxxxx xxx xx xxxxxxxx xxxx xxxxxxxxxxx |

Note: S = Safety Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Criterion Failed.

Listing 16.2.3: Analysis Populations (Page xx of yy)

| Subject | Age/Sex | Parent Study | Population | Included | Reason(s) Excluded |
|---|---|---|---|---|---|
| XXXXXX | XXXX | xxxx | Safety | XXX | |
| xxxxxx | xxxx | XXXX | Safety | xxx | |
| xxxxxx | XXXX | XXXX | Safety | xxx | |
| xxxxxx | XXXX | xxxx | Safety | xx | xxxxxxxxxxxx |

Listing sorted by Subject and Population (as ordered above).

# Listing 16.2.4.1: Subject Demographic Information (Page xx of yy)

| Subject | Evaluable | B: Date of Bir<br>A: Age<br>S: Sex | R: Race<br>E: Ethnicity | Childbearing Potential<br>Method of Contraception | I: Informed Consent Date/Protocol Version P: Did subject consent to photography? |
|---|---|---|---|---|---|
| xxxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxxx | R: xxxxxx xxxxxxxx<br>xx xxxxx xxxxxxx<br>xxxxxx | xxx<br>xxxxxxxxx xxxxxxxxx<br>xxxxxxxxx xxxxxxxx | I: V2.1/xxxx-xx-xx<br>V3/xxxx-xx-xx<br>P: xxx |
| xxxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | xx | I: V2/xxxx-xx-xx<br>P: xxx |
| XXXXXX | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxx | R: xxxxx<br>E: xxxxxxx xx xxxxx | xxx<br>xxxxxxx xxxxxxxxxxxx | I: V3/xxxx-xx-xx<br>P: xxx |

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject. Include all instances of informed consents and associated protocol versions.

# Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Medical History Verbatim Term |
|---|---|---|
| xxxx xxx xxxxx | XXXX XXX XXXXX | xxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |
| xxxx xxx xxxxx | xxxx xxx xxxxx | xxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Medical History Verbatim Term.

# Listing 16.2.4.2.2: Medical History (Page xx of yy)

| Subject | Age/Sex | Evaluable | M: Medical Condition | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | S: Onset Date<br>E: End Date |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | M: xxxx xxxxxxx (xxxxxxx xxxxx) | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxx xxxxxxx | S: xxxx-xx-xx<br>E: |
| | | | M: xxxx xxxxxxx (xxxxxxxx xxxxx) | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxxx xxxxxxx | S: xxxx-xx-xx<br>E: |

Note: S = Safety Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Medical Condition/Surgery Verbatim Term, Onset Date, and End Date.
# Listing 16.2.4.3: Pruritic Disease History (Page xx of yy)

| Subject | Age/Sex | Evaluable | Indication | Date of<br>Diagnosis | Body Locations<br>Affected |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | Prurigo Nodularis | xxxx-xx-xx | xxxxxxxx xxxxx; xxxxxx; xxxx<br>xxx xxxx; xxxxxxxx |
| xxxxxx | xxxx | xxxxxxx | Atopic Dermatitis | xxxx-xx-xx | xxxxxxxx xxxxx; xxxxx xxxxx;<br>xxxxx; xxxxxxxx |

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

Listing 16.2.4.4.1: Unique Medication Names Coded to WHO DDE ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Standardized Medication Name | Medication Name | I: Indication<br>R: Route |
|---|---|---|---|
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |

Note: Standardized Medication Name and ATC Level 2 Term map to the WHO DDE (Version September 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Standardized Medication Name, Medication Name, Indication, and Route.

Note to Programmer: If Indication or Route is 'Other' then the applicable variable is 'OTHER: <specification of other>'.

### Listing 16.2.4.4.2: Concomitant Medications (Page xx of yy)

| | | | M: Medication Name | T: Prior/Concomitant | D: Dose |
|---|---|---|---|---|---|
| | | | P: Standardized Medication Name | F: Date of First Dose | U: Units |
| | | | A: ATC Level 2 Term | S: Start Date (Day) 1 | F: Frequency |
| Subject | Age/Sex | Evaluable | I: Indication | E: End Date (Day) 1 | R: Route |
| xxxxx | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xx |
| | | | P: xxxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx-xx (xx) | F: xxxx |
| | | | I: xxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxx |
| | | | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxxxx |
| | | | P: xxxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx | F: xx |
| | | | I: xxxxxxx | E: | R: xxxx |
| xxxxx | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxx |
| | | | P: xxxxxxxxxxxx | F: xxxx-xx-xx | U: xx |
| | | | A: xxxxxxxxxxx | S: xxxx-xx-xx (x) | F: xx |
| | | | I: xxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxx |

Note to Programmer: If Units, Frequency, Indication, or Route is 'Other' then the applicable variable is 'OTHER: <specification of other>'.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: S = Safety Population.

Standardized Medication Name and ATC Level 2 Term map to the WHO DDE (Version September 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date.

Listing 16.2.4.5: Concomitant Procedures/Therapies (Page xx of yy)

| | | | | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup> | Reason for Procedure |
|---|---|---|---|---|---|
| ubject | Age/Sex | Evaluable | Procedure/Therapy | E: End Date (Day) 1 | or Therapies |
| xxxx | xxxx | xxxxxxxxx | xxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | | S: xxxx-xx-xx (xx) | xxxxxxxx |
| | | | | E: xxxx-xx-xx (xx) | |
| XXXXX | xxxx | xxxxxxxxx | xxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | | S: xxxx-xx | XXXXXXXX |
| | | | | E: xxxx-xx-xx (xx) | |
| XXXX | xxxx | xxxxxxxxx | xxxxxxxxxxx | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | | S: xxxx-xx-xx (xx) | XXXXXXXX |
| | | | | E: xxxx-xx-xx (xx) | |
| | | | | F: xxxx-xx-xx | x xxxxxx xxxx xxxxxx |
| | | | | S: xxxx-xx-xx (xx) | xxxxxxxx |
| | | | | E: xxxx-xx-xx (xx) | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Procedure/Therapy. If ongoing, include 'Ongoing' in place of End Date.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Listing 16.2.4.6: Physical Examination (Page x of xx)

| Subject | Age/Sex | Evaluable | Visit | Date of Assessment (Day) <sup>1</sup> | Physical Exam Completed |
|---|---|---|---|---|---|
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxxx | xxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |
| xxxxxxxx | XXXX | xxxxxxxx | xxxxxxxx | xxxx-xx-xx (x) | xxxxxxx |
| xxxxxxxx | XXXX | xxxxxxxx | xxxxxxxxx | xxxx-xx-xx (xx) | xxxxxx |
| xxxxxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxx-xx-xx (xx) | xxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

### Listing 16.2.5.1: Study Visit Compliance (Page xx of yy)

| Subject | Age/Sex | Evaluable | · Visit | Visit Date | Visit Not Done/<br>Reason for Unscheduled Visit |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xx | |
| | | | xxxxxxx | xxxx-xx-xx | |
| | | | xxxxxx | xxxx-xx-xx | |
| | | | xxxxxx | xxxx-xx-xx | x xxxx xxx xxx xx xxx xxx xxxx xxxxx xxxx |
| | | | xxxxxx | xxxx-xx-xx | |
| | | | xxxxxxxxxxxx | xxxx-xx-xx | |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xx | |
| | | | xxxxx | xxxx-xx-xx | |
| | | | xxxxxxxxxxxx | xxxx-xx-xx | |

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, and Visit Date.

Note to Programmer: If a visit is ranged present the 'Visit Date' column as '<Start Date> to <End Date>' same with the Study Day column.

<sup>1</sup> Day is calculated as date - baseline date for dates prior to baseline date. Otherwise, day is calculated as date - baseline date + 1 for dates on or after baseline date.

Listing 16.2.5.2: Study Drug Dispensing and Return (Page xx of yy)

| Subject | Age/Sex | Evaluable | Bottle<br>Number | Date Bottle<br>Dispensed | Date Bottle<br>Returned | Number of Tablets<br>Dispensed | Number of Tablets<br>Returned | Tablets Used |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx-xx-xx<br>xxxx-xx-xx | xxxx-xx-xx | xx<br>xx | xx<br>xx | xx<br>xx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxx-xx-xx<br>xxxx-xx-xx | xxxx-xx-xx<br>xxxx-xx | xx<br>xx | xx<br>xx | xx<br>xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Date Bottle Dispensed, and Date Bottle Returned.

Listing 16.2.6.1: Worst Itch Numeric Rating Scale (WI-NRS) (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date of Assessment (Day) 1 | WI-NRS <sup>2</sup> in the past 24 hours |
|---|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxxxxx | xxxx-xx-xx (xx) | xx |
| xxxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxxxxxx | xxxx-xx-xx (xx) | xx |
| xxxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxxxxxx | xxxx-xx-xx (xx) | xx |
| xxxxxxx | XXXX | xxxxxxxx | xxxxxxxxxxxxxxxx | xxxx-xx-xx (xx) | xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

 $<sup>^{\</sup>rm 2}$  Scaled from 0 - No Itch to 10 - Worst Itch Imaginable.

### Listing 16.2.6.2: IGA PN-S Results (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date of Assessment (Day) 1 | Investigator's Global Assessement of Prurigo Nodularis Stage |
|---|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxx | xxxx-xx-xx (xx) | xxxxx x |
| | | | xxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |
| | | | xxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |
| | | | xxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |
| | | | XXXXXXXXXXX | xxxx-xx-xx (xx) | XXXXX X |
| | | | XXXXXXXXXXX | xxxx-xx-xx (xx) | xxxxx x |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxxxxxx | xxxx-xx-xx (xx) | xxxxx x |
| | | | xxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |
| | | | xxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |
| | | | XXXXXXXXXXX | xxxx-xx-xx (xx) | XXXXX X |
| | | | XXXXXXXXXXX | xxxx-xx-xx (xx) | XXXXX X |
| | | | xxxxxxxxxxxx | xxxx-xx-xx (xx) | XXXXX X |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.6.3: Dermatology Life Quality Index (DLQI) (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit<br>Date of Assessment | (Day) 1 | Question<br>Number | Question | Result |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxxx | xxxxxxxxx<br>xxx-xx-xx (xx) | | 1 | Over the last week, how itchy, sore, painful or stinging has your skin been? | xxxxxx |
| | | | | | 2 | Over the last week, how embarrassed or self conscious have you been because of your skin? | xxxxxx |
| | | | | | 3 | Over the last week, how much has your skin interfered with you going shopping or looking after your home or garden? | xxxxxx |
| | | | | | 4 | Over the last week, how much has your skin influenced the clothes you wear? | XXXXXX |
| | | | | | 5 | Over the last week, how much has your skin affected any social or leisure activities? | XXXXXX |
| | | | | | 6 | Over the last week, how much has your skin made it difficult for you to do any sport? | XXXXXX |
| | | | | | 7 | Over the last week, has your skin prevented you from working or studying? | XXXXXX |
| | | | | | 7A | If "No", over the last week how much has your skin been a problem at work or studying? | XXXXXX |
| | | | | | 8 | Over the last week, how much has your skin created problems with your partner or any of your close friends or relatives? | xxxxxx |
| | | | | | 9 | Over the last week, how much has your skin caused any sexual difficulties? | XXXXXX |
| | | | | | 10 | Over the last week, how much of a problem has the treatment for your skin been, for example by making your home messy, or by taking up time? | XXXXXX |
| | | | | | | Questionnaire Score | XX |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

# Listing 16.2.6.4: Photography (Page xx of yy)

| Subject | Age/Sex | | Visit<br>Date of Ass | sessment (Day)¹ | Body Areas | s Photographed | d |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxx | xxxxxx | xxxxxxxxx<br>xxx-xx-xx | | xxxxxxx; | xxxxxxxxx; | xxxxxxxx |
| | | | xxxxxxxxx<br>xxx-xx-xx | | xxxxxxx; | xxxxxxxxxx; | xxxxxxxx |
| | | | xxxxxxxxx<br>xxx-xx-xx | | xxxxxxxx; | xxxxxxxxxx; | xxxxxxxx |
| | | | xxxxxxxx<br>xxx-xx-xx | | xxxxxxxx; | xxxxxxxxxx; | xxxxxxxx |

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.1.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| xxxxx xxxxx xxxxx | xxxxx xxxxx xxxxx | xxxxxxxxx |
| | | xxxxxxx xxxxxxx xxxxxxxx |
| | | xxxxxxx xxxxxxxx xxxxxxxxxxxxx |
| | xxxxx xxxxx xxxxx | xxxxxxxxx |
| | | xxxxxxx xxxxxxx xxxxxxxx |
| | | xxxxxxx xxxxxxxx xxxxxxxxxxxxx |
| | xxxxxxxxx | xxxxx xxxxx xxxxx |
| | | xxxxxxx xxxxxxx xxxxxxxx |
| | | xxxxxxx xxxxxxxx xxxxxxxxxxxxx |

Note: System Organ Class and Preferred Term map to MedDRA (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, Preferred Term, and Adverse Event.

#### Listing 16.2.7.1.2: Treatment-Emergent Adverse Events (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | A: Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | S: Grade <sup>2</sup> R: Relationship to Study Treatment O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Action Taken with Study Treatment A: Any Other Action(s) |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (x) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |

Note: S = Safety Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

### Listing 16.2.7.1.3: Serious Adverse Events (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | A: Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup> | S: Grade <sup>2</sup> R: Relationship to Study Treatment O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Action Taken with Study Treatment A: Any Other Action(s) |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| | C: xxxxxxxxxxxxxx | S: $xxxx-xx-xx$ (x) | R: xxxxxxxxxx | R: xxxx xxx xxxxxxx |
| | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxx | R: xxxx xxx xxxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |
| S: xxxxxx | A: xxxxxxxxxxxxxx | F: xxxx-xx-xx | S: xxxx | S: xx |
| A: xxxx | C: xxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | R: xxxxxxxxx | R: xxxx xxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | O: xxxxxxxxx | T: xxx |
| | | | | A: xxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

 $<sup>^2</sup>$  Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death. Note: S = Safety Population.

System Organ Class and Preferred Term map to MedDRA (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.1.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events (Page xx of yy)

| | | Completion/Discontinuation D: Date of Study Discontinuation (Day) 1 | <br> | dverse Events |
|---|---|---|---|---|
| | F: Date of First | T: Primary Reason for Treatment | A: Event | S: Start Date (Day) 1 |
| S: Subject | Dose | Discontinuation | S: Grade <sup>2</sup> | E: End Date (Day) 1 |
| A: Age/Sex | L: Date of Last | S: Primary Reason for Study | R: Relationship to | A: Action Taken with Study |
| E: Evaluable | Dose | Discontinuation | Study Treatment | Treatment |
| S: xxxxxx | F: xxxx-xx-xx | D: xxxx-xx-xx (xx) | A: xxxxxxxxx | S: xxxx-xx-xx (xx) |
| A: xxxx | L: xxxx-xx-xx | T: xxxxxx | S: xxxxxxx | E: xxxx-xx-xx (xx) |
| E: xxxxxxx | | S: xxxxxxxxxxxxx | R: xxxxxxxxxxxxxxx | A: xxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death.

#### Listing 16.2.7.2.1: Hospital Anxiety and Depression Scale (Page xx of yy)

V: Visit Subject Age/Sex Evaluable D: Date of Assessment (Day) 1 Question Result XXXXXXXX XXXX xxxxxxx V: xxxxxxxxx I feel tense or 'wound up' XXXXXXXXXXXXXXXXX I still enjoy the things I used to enjoy D: xxxx-xx-xx (xx) xxxxxxxxxxxxxxxxx I get a sort of frightened feeling as if something awful is about to happen XXXXXXXXXXXXXXXXXX I can laugh and see the funny side of things XXXXXXXXXXXXXXXXX Worrying thoughts go through my mind XXXXXXXXXXXXXXXXX I feel cheerful xxxxxxxxxxxxxxx I can sit at ease and feel relaxed xxxxxxxxxxxxxxxxxxxxxDepression Subscale Anxiety Subscale XX

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.

#### Listing 16.2.7.2.2: Epworth Sleepiness Scale (Page xx of yy)

V: Visit Subject Age/Sex Evaluable D: Date of Assessment (Day) 1 Situation Result XXXXXXXX XXXX xxxxxxx V: xxxxxxxxx Sitting and reading XXXXXXXXXXXXXXXXXX D: xxxx-xx-xx (xx) Watching TV xxxxxxxxxxxxxxxxx Sitting, inactive in a public place (e.g. a theatre or a meeting) XXXXXXXXXXXXXXXXXX As a passenger in a car for an hour without a break XXXXXXXXXXXXXXXXX Lying down to rest in the afternoon when circumstances permit xxxxxxxxxxxxxxxxx Sitting and talking to someone XXXXXXXXXXXXXXXXXX Sitting quietly after a lunch without alcohol XXXXXXXXXXXXXXXXXX In a car, while stopped for a few minutes in the traffic XXXXXXXXXXXXXXXXXX

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

# Listing 16.2.7.3: Menstrual Diary (Page xx of yy)

| Subject Age/Sex Evaluable | Childbearing Potential | Start Date of Period (Day)¹ | End Date of Period (Day) 1 |
|---|---|---|---|
| xxxxxxx xxxx xxxxx | xxxxxxxxxxx | xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx) | xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx)<br>xxxx-xx-xx (xx) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.

Listing 16.2.8.1: Pregnancy Test Results (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | V: Visit<br>D: Date (Day) <sup>1</sup> | S: Specimen <sup>2</sup><br>R: Result | S: Was a Serum Pregnancy Test Ordered? E: If no, but was required, explain | Comments |
|---|---|---|---|---|
| S: xxxxxx | V: xxxxxxxx | S: xxxxx | S: xxx | xxxxxxxxxxx |
| A: xxxx<br>E: xxxxxxxx | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| | V: xxxxxxxx | S: xxxxx | S: xx | |
| | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: | |
| S: xxxxxx | V: xxxxxxxx | S: xxxxx | S: xx | |
| A: xxxx<br>E: xxxxxxx | D: xxxx-xx-xx (xxx) | R: xxxxxxxx | E: xxxxxxxxxxxxxxxxxxxxxxxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Specimen. NOTE: Serum Pregnancy Questions (S: E:) are only applicable to Urine Pregnancy test records.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> For Serum pregnancy results: HCG levels less than 10 mIU/mL are considered negative for pregnancy. Levels between 10 - 24.9 mIU/mL are equivocal and a redraw of the patient after 48 hours is suggested. Levels greater than or equal to 25 mUI/mL are considered positive for pregnancy.

## Listing 16.2.8.2.1: Laboratory Test Results (Page xx of yy)

| _ | V: Visit D: Date (Day) 1 C: Category | Laboratory Test | Results<br>(Units) | Low | | rence Range<br>Indicator | Comments |
|---|---|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx (xxx)<br>C: xxxxxxxxxxxxxxxxxxxxx | ******* | xxxx (xxxxxx) | | | | ************************************** |
| | V: xxxxxxxxx D: xxxx-xx-xxTxx:xx:xx (xxx) C: xxxxxxxxxxxxxxxxxxxx | ********** | xxxx (xxxxxx) | Х | xx | xxxxxxxxxx (xx | x) xxxxxxxxxxxxx<br>xxxxxxxxxxxxxxx<br>xxxxxxxx |
| | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx (xxx)<br>C: xxxxxxxxxxxxxxxxxxxxx | ***** | xxxx (xxxxxx) | Х | XX | xxxxxxxxxx (xx | х) |

Note: S = Safety Population.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Category, and Lab Test.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

### Listing 16.2.8.2.2: Out of Range Laboratory Results (Page xx of yy)

| - | V: Visit D: Date (Day) 1 e C: Category | Laboratory Test | Results<br>(Units) | Low | | rence Range_<br>Indicator(CS²) | Comments |
|---|---|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx (xxx)<br>C: xxxxxxxxxxxxxxxxxxxx | ******* | xxxx (xxxxxx) | | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | V: xxxxxxxxx D: xxxx-xx-xxTxx:xx:xx (xxx) C: xxxxxxxxxxxxxxxxxxxxx | ******** | xxxx (xxxxxx) | х | XX | xxxxxxxxx (xxx) | ************************************** |
| | V: xxxxxxxxx D: xxxx-xx-xxTxx:xx:xx (xxx) C: xxxxxxxxxxxxxxxxxxxx | ***** | xxxx (xxxxxx) | Х | xx | xxxxxxxxxx (xxx) | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Category, and Lab Test.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

 $<sup>^2</sup>$  Clinical significance based on Investigator interpretation. CS = Clinically Significant; NCS = Not Clinically Significant. Note: S = Safety Population.

## Listing 16.2.8.2.3: Laboratory Information Captured within Case Report Forms (Page xx of yy)

| S: Subject<br>A: Age/Sex | | Y: Was sample collected? | |
|---|---|---|---|
| E: Evaluable | e C: Category | D: Date of Sample Collection | Were there any abnormal results? |
| S: xxxxxx | V: xxxxxxxx | Y: xxx | |
| A: xxxx<br>E: xxxxxxx | C: xxxxxxxxxxxxxxxxxxxx | D: xxxx-xx-xx | xxxxxxxxxxxx |
| S: xxxxxx | V: xxxxxxxx | Y: xxx | |
| A: xxxx<br>E: xxxxxxx | C: xxxxxxxxxxxxxxxxxxxx | D: xxxx-xx-xx | xxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, Category, and Lab Test.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: S = Safety Population.

Listing 16.2.8.2.4: Common Laboratory Comments Including Reference Ranges for Specific Laboratory Tests (Page 1 of 1)

| Category | Laboratory Test | Comments |
|---|---|---|
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | *************************************** |
| | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ***************************** |
| | | *************************************** |
| | | ************************* |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ***************************** |
| | | *************************************** |
| | | *************************************** |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx | *************************************** |
| | | ***************************** |
| | | *************************************** |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Category and Lab Test.

#### Listing 16.2.8.3: Electrocardiogram Test Results (Page x of xx)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | Category | ECG Parameter | V: Visit<br>D: Date/Time of ECG (Day) <sup>1</sup> | Result (unit) | Clinical<br>Significance <sup>2</sup> | Comments |
|---|---|---|---|---|---|---|
| S: xxxxxxxx<br>A: xxxx<br>E: xxx/xx/xxx | xxxxxxxx | xxxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx (xx) | xxxx xxxxx xx (xxx) | xxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Category, Parameter, Visit, and Date. Note: for interpretation records, EGEVAL should be concatenated into ECG Parameter as EGTEST (EGEVAL).

Include information captured within CRF as a separate parameter within listing.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

 $<sup>^2</sup>$  Clinical significance based on Investigator interpretation. CS = Clinically Significant; NCS = Not Clinically Significant. Note: S = Safety Population.

Listing 16.2.8.4: Vital Signs (Page x of xx)

| Subject | Age/Sex | Evaluable | Visit | Date of Measurements (Day) $^{\mathrm{1}}$ | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| xxxxxxxx | xxxx | xxxxx | xxxxxxxxx | xxxx-xx-xx (xxx) | xxxxx xxx | xx | xxxx |
| | | | | , | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | XX | xxxx |
| | | | XXXXX XXX | xx | xxxx | | |
| | xxxxxxxxx | xxxx-xx-xx (xxx) | xxxxx xxx | xx | xxxx | | |
| | | | | xxxxx xxx | XX | XXXX | |
| | | | xxxxx xxx | XX | XXXX | | |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| xxxxxxx | XXXX | xxxxx | xxxxxxxx | xxxx-xx-xx (xxx) | XXXXX XXX | XX | xxxx |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | xxxxxxxxx | xxxx-xx-xx (xxx) | xxxxx xxx | XX | xxxx |
| | | | | | xxxxx xxx | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |
| | | | | | XXXXX XXX | XX | XXXX |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date, and Vital Sign (ordered as: Height, Weight, Temperature, Respiration Rate, Heart Rate, Systolic Blood Pressure, Diastolic Blood Pressure).